CLINICAL TRIAL: NCT07130201
Title: Sleep Disorders and Automatic Dysfunction in Elderly Cardiovascular Patients: Risk Factors and Clinical Implications "
Brief Title: Sleep and Automatic Dysfunction in Elderly Cardiovascular Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa sedek Roshdy, Principal Investigator, Assiut University
Other Study IDs: SD_AD_ECP
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Study group: Patients with cardiovascular diseases

SUMMARY:
This study explores the relationship between sleep disorders and autonomic dysfunction in elderly patients with cardiovascular disease. It examines common risk factors such as aging-related physiological changes, comorbidities, and lifestyle factors, and discusses how disturbances in sleep and autonomic regulation can worsen cardiovascular outcomes. The work also outlines potential clinical implications, including the importance of early screening, integrated management strategies, and targeted interventions to improve both cardiovascular health and quality of life in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

- Patients will be recruited from the outpatient clinic (to include stable patients) Age ≥ 65 years Clinically diagnosed cardiovascular disease (e.g., heart failure, atrial fibrillation, coronary artery disease) Able to provide informed consent

Exclusion criteria:

Diagnosed neurodegenerative diseases (e.g., advanced dementia) Use of sedatives/hypnotics in the past 2 weeks Terminal illness or palliative care status

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with cardiovascular diseases more than 65 years old
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disturbance | Baseline
  Prevalence of sleep disturbance among elderly patients with cardiovascular diseases